CLINICAL TRIAL: NCT02964455
Title: A Prospective, Open-label, Phase I Study of Docetaxel and Nedaplatin Twice Weekly in Combination With Chest Radiotherapy in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Study of Concurrent Chemoradiotherapy for Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO201610003
Record Dates: First submitted 2016-11-13; First posted 2016-11-16 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Chemoradiotherapy; Docetaxel; Nedaplatin; Twice weekly
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel + Nedaplatin + Radiotherapy (Experimental): Docetaxel and nedaplatin 5 mg/m², 10 mg/m², or 15 mg/m² given intravenously twice weekly (depending on dose under investigation at time of registration) on days 1,4 (depending on allocation of treatment schedule) for 4-6 weeks during chest radiation.
  Interventions: Drug: Docetaxel; Drug: Nedaplatin; Radiation: chest radiation

INTERVENTIONS:
Drug: Docetaxel — 5 mg/m², 10 mg/m², or 15 mg/m² given intravenously twice weekly (depending on dose under investigation at time of registration) on days 1,4 (depending on allocation of treatment schedule) for 4-6 weeks during chest radiation
Drug: Nedaplatin — 5 mg/m², 10 mg/m², or 15 mg/m² given intravenously twice weekly (depending on dose under investigation at time of registration) on days 1,4 (depending on allocation of treatment schedule) for 4-6 weeks during chest radiation
Radiation: chest radiation — continuous chest radiation at 64 Gy/32f

SUMMARY:
The phase I study is to determine the maximum tolerated dose and dose limiting toxicity of docetaxel and nedaplatin prescribed twice weekly in combination with concurrent chest radiotherapy in patients with locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma
* Inoperable stage II-III (AJCC/UICC; seventh edition), confirmed by contrast- enhanced computed tomography,endoscopic ultrasonography, barium esophagram, emission computed tomography and/or positron emission tomography/computed tomography.
* Eastern Cooperative Oncology Group (ECOG) performance status 1-2
* Estimated life expectancy of at least 12 weeks
* Charlson comorbidity index≤4
* Adequate bone marrow function: white blood cells grade 0 or 1,absolute neutrophils grade 0 or 1, platelets grade 0, haemoglobin grade 0 or 1
* Adequate renal function: creatinine grade 0 or 1
* Adequate liver function: serum bilirubin grade 0 or 1, alanine aminotransferase and aspartate aminotransferase <2 times of the upper normal limit
* Weight loss≤15% during 6 months prior to diagnosis
* Forced expiratory volume second≥1L

Exclusion Criteria:

* Prior history of malignancy, except for nonmelanoma skin carcinoma or cervical carcinoma in situ
* Previous anti-tumor therapy, including surgery, chemotherapy or radiotherapy
* Contraindication for chemotherapy or radiotherapy
* Malignant pleural or pericardial effusion
* Women in pregnancy or lactation period
* Women who has the probability of pregnancy without contraception
* Weight loss≥15% during 3 months prior to diagnosis
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity | From start of week 1 to 2 weeks after end of combination treatment (combination treatment = 6.5 weeks)
Maximum tolerated dose | From start of week 1 to 2 weeks after end of combination treatment (combination treatment = 6.5 weeks)

SECONDARY OUTCOMES:
Occurrence and severity of adverse events | From start of week 1 to 6 weeks after end of combination treatment (combination treatment = 6.5 weeks)
Clinical response rate | 8 weeks after end of combination treatment
Dynamic plasma concentration of docetaxel and nedaplatin | From start of week 1 to the end of combination treatment (6.5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Prof., Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No